CLINICAL TRIAL: NCT05814471
Title: Protocol for the Clinical Validation of a Valgus Knee Brace for Gonarthrosis
Brief Title: Validation of a Knee Brace for Gonarthrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TOPMED (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other); Laboratoire Victhom (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RD-241-VicD_1
Record Dates: First submitted 2023-03-16; First posted 2023-04-14 (Actual); Results first posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Gonarthrosis
Keywords: knee brace; orthosis; treatment efficacy; arthrosis; comfort; ease of use
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Randomized trial with condition crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adjustement period(velcro)first, then Cable fastening system then Velcro Straps (Experimental): A new knee brace is worn for a 14 days adjustement period with velcro straps. Then the brace is worn with a cable fastening system for a first 14 days intervention period, therefore the knee brace is held in place by a cable fastening system and 3d printed straps. The second 14 days intervention period is done with velcro straps keeping the brace in position.
  Interventions: Device: Cable fastening system and 3d printed straps(14 days); Device: Velcro straps system(14 days); Device: Adjustment period(Velcro-14 days)
- Adjustement period(velcro)first, then Velcro Straps then Cable fastening system (Active Comparator): A new knee brace is worn for a 14 days adjustement period with velcro straps. The first 14 days intervention period is done with velcro straps keeping the brace in position. Then the brace is worn with a cable fastening system for a second 14 days intervention period, therefore the knee brace is held in place by a cable fastening system and 3d printed straps.
  Interventions: Device: Cable fastening system and 3d printed straps(14 days); Device: Velcro straps system(14 days); Device: Adjustment period(Velcro-14 days)

INTERVENTIONS:
Device: Cable fastening system and 3d printed straps(14 days) — The participants will wear a Odra knee brace held in place with by a cable fastening system and 3d printed straps for 2 weeks.
Device: Velcro straps system(14 days) — The participants will wear a Odra knee brace held in place with by a velcro straps system for 2 weeks.
Device: Adjustment period(Velcro-14 days) — The participants will wear a new Odra knee brace held in place with by a velcro straps system for 2 weeks.

SUMMARY:
A study about the effects of different fastening systems for knee braces on comfort, ease of installation and treatment efficacy both physical and psychological. Two different systems will be tested, velcro straps and a cable-fastening system.

DETAILED DESCRIPTION:
There are 2 main types of knee braces for gonarthrosis: soft knee braces and rigid knee braces. Soft knee braces use malleable materials such as cloth or rubber to apply forces on the leg whereas rigid braces use plastic or metal shells. Three main types of fastening systems are used on these types of orthoses: velcro systems, hybrid systems and cable fastening systems. Therefore, different configurations exist to reduce biomechanical deficits caused by the pathology.

Each fastening system has its advantages and disadvantages. Velcro straps are fast and intuitive to use, altough multiple difficulties are mentionned: adjusment, cleaning, the number of straps needed to maintain the knee brace in position as well as the noise while detaching the straps. Hybrid systems regularly use velcro straps to which are added quick-release fasteners to simplify the installation and uninstallation process. Cable fastening systems also use quick-release fasteners. The adjusment process is simple and precise with minimal noise with these systems.

Comfort, efficacy and ease of use are essential qualities of a knee brace. Confort is primordial as it is directly linked to treatment adherence by the patients. Efficacy of a knee brace treatment may be measured by symptom or medication use evolution but also with daily practice of problematic movement by the patient. Ease of use must be optimized as it presents an opportunity to increase treatment adherence. The goal of the fastening system developped in partnership with Laboratoires Victhom is to increase ease of use of the knee brace while maintaining comfort and treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Has worn an ODRA knee brace multiple hours a day during the last 6 months

Exclusion Criteria:

* Wounds on the lower body

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2025-01-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- TOPMED, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total enrollment was 5 participants, since participants did all interventions in a sequence, the total amount of participants for each intervention was 5 since there were no exclusions nor drop-outs.
Period: Adjustment Period(14 Days)
Arm/Group | Adjustement Period(Velcro)First, Then Cable Fastening System Then Velcro Straps | Adjustement Period(Velcro)First, Then Velcro Straps Then Cable Fastening System
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0
Period: First Intervention(14 Days)
Arm/Group | Adjustement Period(Velcro)First, Then Cable Fastening System Then Velcro Straps | Adjustement Period(Velcro)First, Then Velcro Straps Then Cable Fastening System
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0
Period: Second Intervention(14 Days)
Arm/Group | Adjustement Period(Velcro)First, Then Cable Fastening System Then Velcro Straps | Adjustement Period(Velcro)First, Then Velcro Straps Then Cable Fastening System
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants who completed the intervention protocol.
Arm/Group | All Participants
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  Canada | 5
Psychological Symptoms [Mean (Standard Deviation); unit: units on a scale] — Psychological Symptoms Inventory Total Score(Ilfeld, F. W. (1976). Further validation of a psychiatric symptom index in a normal population. Psychological Reports, 39(3, Pt 2), 1215-1228.). Total scores ranges from 0 (no symptoms) to 100 (high levels of anxiety, depression hostility and concentration symptoms).
  units on a scale | 28.0 (27.4)
Physical Symptoms [Mean (Standard Deviation); unit: units on a scale] — Knee injury and Osteoarthritis Outcome Total Score (KOOS), translated to French(Quebec). Total scores ranges from 0 (extreme knee problems) to 100 (no symptoms).
  units on a scale | 68.9 (23.9)

OUTCOME MEASURES:

1. Primary Outcome: Ease of Use Measurement Scale
Description: The scale was developped for this study. The mesure is an average of 5 items with 5 point scale rating system(1 harder to use; 5 easier to use). Mean score ranges from (1 harder to use; 5 easier to use)
Time Frame: Before the 2 weeks of intervention with each brace, assessed after a brace fitting protocol and a few minutes of wearing the intervention brace.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Cable Fastening System: The knee brace is worn for 2 weeks after adjustment period. The knee brace is held in place by a cable fastening system and 3d printed straps.
  Cable fastening system and 3d printed straps: The participants will wear a Odra knee brace held in place with by a cable fastening system and 3d printed straps for 2 weeks.
- Velcro Straps: The knee brace is worn for 2 weeks after adjustment period. The knee brace is held in place by a velcro straps system.
  Velcro straps system: The participants will wear a Odra knee brace held in place with by a velcro straps system for 2 weeks.
- Adjustment Period(Velcro-14 Days): The participants wore a new Odra knee brace held in place with by a velcro straps system for 2 weeks.
Arm/Group | Cable Fastening System | Velcro Straps | Adjustment Period(Velcro-14 Days)
Number analyzed (Participants) | 5 | 5 | 5
score on a scale | 4.05 (0.26) | 3.00 (1.21) | 4.05 (0.78)

2. Primary Outcome: Ease of Use Measurement Scale
Description: as for outcome 1
Time Frame: Directly after the 2 weeks of intervention with each brace, assessed after a brace fitting protocol and a few minutes of wearing the intervention brace.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cable Fastening System | Velcro Straps | Adjustment Period(Velcro-14 Days)
Number analyzed (Participants) | 5 | 5 | 5
score on a scale | 4.60 (0.33) | 3.45 (1.17) | 3.80 (0.54)

3. Primary Outcome: Comfort Measurement Scale
Description: The scale was developped for this study. The mesure is an average of 2 items with 5 point scale rating system(1 lowest comfort; 5 highest comfort). Total score is adjusted to 0 (lowest comfort) to 100 (highest comfort).
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cable Fastening System | Velcro Straps | Adjustment Period(Velcro-14 Days)
Number analyzed (Participants) | 5 | 5 | 5
score on a scale | 90 (13.7) | 80 (20.9) | 62.5 (20.9)

4. Primary Outcome: Comfort Measurement Scale
Description: as for outcome 3
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cable Fastening System | Velcro Straps | Adjustment Period(Velcro-14 Days)
Number analyzed (Participants) | 5 | 5 | 5
score on a scale | 90 (11.2) | 75 (30.6) | 77.5 (16)

5. Primary Outcome: Physical Symptoms
Description: Knee injury and Osteoarthritis Outcome Total Score (KOOS), translated to French(Quebec). Minimum=0(worst symptoms); Maximum=100(no symptoms);
Time Frame: Change between baseline(directly before adjustment period) and directly after 2 weeks adjustment period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 5
score on a scale | 0.6 (3.6)

6. Primary Outcome: Physical Symptoms
Description: as for outcome 5
Time Frame: Change between directly after 2 weeks adjustment period and directly after 2 weeks of use for each arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cable Fastening System | Velcro Straps
Number analyzed (Participants) | 5 | 5
score on a scale | 2.0 (2.3) | -0.2 (5.4)

7. Primary Outcome: Psychological Symptoms
Description: Psychological Symptoms Inventory Total Score(Ilfeld, F. W. (1976). Further validation of a psychiatric symptom index in a normal population. Psychological Reports, 39(3, Pt 2), 1215-1228.). Minimum=0; (No symptoms); Maximum=100(Worst Symptoms);
Time Frame: Change between baseline(directly before adjustment period) and directly after 2 weeks adjustment period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 5
score on a scale | -3.4 (6.5)

8. Primary Outcome: Psychological Symptoms
Description: as for outcome 7
Time Frame: Change between directly after 2 weeks adjustment period and directly after 2 weeks of use for each arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cable Fastening System | Velcro Straps
Number analyzed (Participants) | 5 | 5
score on a scale | -7.4 (6.1) | -6.7 (6.1)

ADVERSE EVENTS:
Time Frame: 6 weeks (2 weeks adjustment period + 2 weeks of treatment for each arm)
Groups:
- Adjustment Period: The participants will wear a new Odra knee brace held in place with by a velcro straps system for 2 weeks.
Arm/Group | Cable Fastening System | Velcro Straps | Adjustment Period
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is 1 year from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2025-06-25): https://cdn.clinicaltrials.gov/large-docs/71/NCT05814471/Prot_000.pdf
  • Informed Consent Form (2025-06-25): https://cdn.clinicaltrials.gov/large-docs/71/NCT05814471/ICF_001.pdf